CLINICAL TRIAL: NCT03263208
Title: A Study of CD19 CAR-T Cells for Patients With Relapse and Refractory CD19+ B-cell Acute Lymphoblastic Leukemia
Brief Title: CD19 CAR-T Cells for Patients With Relapse and Refractory CD19+ B-ALL.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: The Pregene (ShenZhen) Biotechnology Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HenanCH152
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-08

CONDITIONS: B-cell Acute Lymphocytic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19 CAR-T (Experimental): A conditioning chemotherapy regiment of fludarabine and cyclophosphamide will be administered followed by a single infusion of CAR transduced autologous T cells administered intravenously.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: CD19 CAR-T

INTERVENTIONS:
Drug: Cyclophosphamide — patients will receive a standard pre-conditioning regime with cyclophosphamide 0.6-0.8g/m2/day IV for 2 days(Day-5 to day-4).
Drug: Fludarabine — Fludarabine 25-30mg/m2/day IV for 3 days(Day-5 to day-3).
Biological: CD19 CAR-T — CD19 CAR-T cells will be administered after completion of the chemotherapy.

SUMMARY:
The purpose of this study is to infusion CD19 CAR-T cells to the patients with relapsed and refractory CD19+ B cell leukemia, to assess the safety and feasibility of this strategy. The CAR enables the T cell to recognize and kill the leukemic cell through the recognition of CD19, a protein expressed of the surface of the leukemic cell in patients with CD19+ leukemia.

DETAILED DESCRIPTION:
Upon meeting the eligibility requirements and enrolling on study, Subjects will be collected large numbers of peripheral blood mononuclear cells (PBMC) for the generation of the CD19 CAR-T cells. The T cells are isolated from the PBMC, transduced with a lentivirus to express the CD19 CAR as well as a truncated EGFR that has no signaling capacity (noted EGFRt) and expanded in vitro and then administered to subjects.

Subjects will have blood tests to assess safety and efficacy, and persistence of the CD19 CAR-T cells on week 4 after their last infusion. Following the 6 months of intensive follow-up, subjects will be evaluated every 10 weeks for 1 year with a physical examination, blood tests, bone marrow aspirate, MRD and persistence of CD19 CAR-T.

Some subjects will receive cetuximab for ablation of the genetically modified T cells. Criteria to receive cetuximab include acute toxicities that are life threatening.

ELIGIBILITY:
Inclusion Criteria:

* 1. 2 years to 70 years, expected survival > 3 months;
* 2. CD19 positive B-cell acute lymphoblastic leukemia;
* 3. ECOG < 2；
* 4. The tumor load in the bone marrow is less than 60%;
* 5. Cardiac function: 1-2 levels; Liver: TBIL≤3ULN，AST ≤2.5ULN，ALT ≤2.5ULN; kidney: Cr≤1.25ULN; Peripheral Blood: WBC ≥ 2.0×109/L, Hb ≥80 g/L, PLT ≥ 30×109/L）;
* 6. No leukemia cells in the central nervous system;
* 7. No serious allergic constitution;
* 8. No other serous diseases that conflicts with the clinical program;
* 9. No other cancer history;
* 10. No serious mental disorder;
* 11. female participants of reproductive potential must have a negative serum pregnancy test;
* 12. Informed consent is signed by a subject or his lineal relation.

Exclusion Criteria:

* 1. Pregnant or lactating women;
* 2. Uncontrolled active infection, HIV infection, syphilis serology reaction positive;
* 3. Active hepatitis B or hepatitis C infection;
* 4. Recent or current use of glucocorticoid or other immunosuppressor;
* 5. With severe cardiac, liver, renal insufficiency, diabetes and other diseases;
* 6. Participate in other clinical research in the past three months; previously treatment with any gene therapy products;

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-08-16 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
safety as assessed by the occurence of study related adverse events | 30 days
  number of participants with adverse events
anti-tumor responses of CD19 CAR-T cells | 1 year

SECONDARY OUTCOMES:
Persistence of the CD19 CAR+ T cells | 1 year
  determine duration of in vivo survival of CD19 CAR-T cells
Number of participants who have T cells ablated with cetuximab | 1 year
  The efficacy of cetuximab to ablate the T cells will be measured by loss of detection of T cells and any associated toxicities as well as facilitating B cell recovery.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan